CLINICAL TRIAL: NCT03770026
Title: Intrauterine Infusion of Autologous Platelet-rich Plasma to Prevent a Thin Endometrium in Infertile Women Undergoing Clomiphene Citrate Therapy: a Pilot Prospective Self-controlled Trial
Brief Title: Autologous Platelet-rich Plasma for Clomiphene Citrate-induced Thin Endometrium
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Professor of Obestetrics and Gynecology, Benha University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 181210
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Infertility, Female, Associated With Anovulation
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clomiphene citrate only (Active Comparator): Infertile women (30 women) with prior clomiphene citrate failure (ovulation was documented without conception), with thin endometrium (<7mm) in at least 3 cycles. Saline cervical flushing will be done at cycle day 8 and 10 to convince patient-blinded procedure.
  Interventions: Drug: clomiphene citrate; Drug: Saline cervical flushing
- Platelet-rich plasma plus Clomiphene (Experimental): Women who did not conceive on the Clomiphene citrate-only cycle will receive Clomiphene citrate 100 mg/ day starting from the third day of the cycle. Intrauterine Autologous platelet-rich plasma will be done on the cycle days 8 and 10.
  Interventions: Drug: clomiphene citrate; Biological: Intrauterine Autologous platelet-rich plasma

INTERVENTIONS:
Drug: clomiphene citrate — Clomiphene citrate-only arm: Patients will receive Clomiphene citrate induction (in a dose of 100 mg/day starting from day 3 of the cycle for 5 days). Sonographic assessment of endometrial thickness together with Power Doppler evaluation endometrial and sub-endometrial blood flow a will be done in the Day of HCG injection.
  Other Names: Clomiphene
Drug: Saline cervical flushing — Cervical irrigation with 1 ml of 0.9% normal saline will be done at cycle day 8 and 10 to convince patient-blinded procedure.
  Other Names: Saline
  Arms: Clomiphene citrate only
Biological: Intrauterine Autologous platelet-rich plasma — Under complete aseptic cares and ultrasound supervision, Autologous platelet-rich plasma (0.5 - 1 ml) was immediately injected into the uterine cavity using an intrauterine insemination catheter in the cycle days 8 and 10. The Autologous platelet-rich plasma is prepared in collaboration with the Department of Clinical Pathology, Faculty of Medicine, Benha University.
  Other Names: Platelet-rich plasma
  Arms: Platelet-rich plasma plus Clomiphene

SUMMARY:
This is a prospective self-controlled clinical study. Women with clomiphene Citrate failure with thin endometrium less than 7 millimeters for at least 3 cycles will be selected (N = 30). Patients will receive 2 ovarian stimulation cycles with Clomiphene citrate (CC) 100 mg/ day for 5 days from cycle day 3. A control cycle (CC only cycle) woman will continue on CC alone plus cervical irrigation of cervix with 1 ml of 0.9% normal saline at cycle day 8 and 10 to assure patient-blinded method. The study group, the same will be done plus the intrauterine infusion of Autologous platelet-rich plasma (PRP) in 8th and 10th days of the cycle. In both groups, the endometrial thickness and Power Doppler evaluation of their endometrial and sub-endometrial blood flow will be measured on the day of Human Chorionic Gonadotropin (HCG) administration.

DETAILED DESCRIPTION:
This is a pilot prospective self-controlled clinical trial. Women with Clomiphene Citrate failure with documented thin endometrium less than 7 millimeters for at least 3 stimulation cycles will be chosen (N = 30). Patients will experience 2 ovarian stimulation cycles with Clomiphene citrate (CC) in a dose of 100 mg/ day for 5 days starting from cycle day 3. A control cycle (CC only cycle) woman will continue on Clomiphene Citrate alone plus cervical irrigation of cervix with 1 ml of 0.9% normal saline at cycle day 8 and 10 to confirm patient-blinded process.

The study group, the same will be done in addition to the intrauterine infusion of with Autologous platelet-rich plasma (PRP) in 8th and 10th days of the cycle.

In both groups, the endometrial thickness and Power Doppler evaluation of their endometrial and sub-endometrial blood flow will be measured on the day of HCG administration.

ELIGIBILITY:
Inclusion Criteria:

* Women with clomiphene citrate failure (defined as at least previous 3 ovulatory cycles with clomiphene citrate, with no pregnancy),
* persistently thin endometrium (less than 7 millimeters in at least 3 cycles).
* normal baseline Follicle Stimulating Hormone, Luteinizing Hormone, and free testosterone levels, patent tubes by hysterosalpingography, and satisfactory male semen analysis

Exclusion Criteria:

* previous ovarian surgery;
* endocrine disorders ;
* pelvic pathologies;
* chronic hepatic, cardiovascular, or renal disease;
* other factors of infertility and
* use of gonadotropins or hormonal contraception through the latest 6 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | 1 day
  Transvaginal sonographic estimation of maximal distance traversing endometrial- myometrial interphase on each endometrial stripe in a -midsagittal plane in the uterine fundus.

SECONDARY OUTCOMES:
Power Doppler estimation of endometrial and sub-endometrial vascularity | 1 day
  Endometrial and sub-endometrial vascularity signals will be evaluated using the power Doppler.
Clinical pregnancy rate | At the end of a 28-day menstrual cycle.
  Recognizing pregnancy through positive urinary HCG test plus sonographic detection of cardiac pulsations

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Walid A Morad, Principal Investigator — Banha Faculty of Medicine, Banha Univerisity
Locations (1):
- Banha Faculty Hospital, Banhā, Alkalubia, Egypt